CLINICAL TRIAL: NCT00534443
Title: A Clinical Study of the Efficacy of Esomeprazole or Rabeprazole on the Pattern of Release of Pro- and Anti-inflammatory Cytokines From Gastric Mucosa of Patients With Peptic Ulcer Disease
Brief Title: Importance of Cytokines in Peptic Ulcer Disease: Implications for Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Evangelos Giamarellos-Bourboulis, University of Athens, Medical School, Greece
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3530
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2008-06

CONDITIONS: Peptic Ulcer
Keywords: peptic ulcer; gastritis; sTREM-1; cytokines; Changes of inflammatory status in gastric mucosa; sTREM-1 as a disease marker
MeSH Terms: conditions — Peptic Ulcer; Gastritis | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): A total of 130 patients with peptic ulcer disease and /or chronic gastritis will be enrolled in the study after written informed consent. Patients will be prescribed oral treatment with rabeprazole or esomeprazole according to standard guidelines. Rabeprazole is administered 20mg twice daily and esomeprazole 10 mg once daily. Selection of rabeprazole or esomeprazole is at the discretion of the attending physicians. The drug is administered for four weeks in patients with duodenal ulcers, for eight weeks in patients with gastric ulcers and for four weeks in patients with chronic gastritis.
  Interventions: Procedure: Endoscopy of upper GI tract

INTERVENTIONS:
Procedure: Endoscopy of upper GI tract — Upper GI endoscopy, one time on diagnosis and a second time 15 days after the end of the treatment. Gastric juice will be aspirated immediately after the entrance of the endoscope into the gastric lumen. Four biopsy specimens will be obtained from adjacent areas of the gastric antrum. Each biopsy will be used for in vitro culture. Blood will be sampled from one antecubital vein under aseptic conditions.
  Each patient will be given antisecretory treatment and - if necessary- eradication treatment of H. pylori according to international guidelines.
  Other Names: Gastroscopy

SUMMARY:
Although all PPIs are effective, there are some differences in their clinical performance, particularly in terms of the degree and speed of gastric acid suppression. Few data are also available about their effect of the pathophysiological mechanisms of gastritis and peptic ulcer disease. Aim of the present study is to investigate the effect of therapy with esomeprazole or rabeprazole on the mechanism of pathogenesis of gastritis and particularly on the pattern of release of pro- and anti- inflammatory cytokines associated to peptic ulcerative process by the gastric mucosa.

DETAILED DESCRIPTION:
Although all PPIs are effective, there are some differences in their clinical performance, particularly in terms of the degree and speed of gastric acid suppression. Few data are also available about their effect of the pathophysiological mechanisms of gastritis and peptic ulcer disease.

Triggering receptor expressed on myeloid cells (TREM)-1 is a recently discovered receptor expressed on the surface of neutrophils and monocytes. Engagement of TREM-1 has been reported to trigger the synthesis of proinflammatory cytokines. A soluble form of TREM-1, named sTREM-1, was observed and identified at significant levels in serum samples from patients with disease of the gastrointestinal tract inflammatory bowel disease. rendering interest about the implication of sTREM-1 in their pathogenesis.

sTREM-1 was also found elevated in the gastric juice of patients with peptic ulcer disease being correlated to the degree of the infiltration of the gastric mucosa by neutrophils.

Published data of our group elicit that sTREM-1 secretion is a crucial parameter for evolution from chronic gastritis to peptic ulcer disease. Samples of biopsies of gastric mucosa were cultured in the absence/presence of endotoxins showing that the inflamed mucosa was a potent secretor of sTREM-1 whatever ceased to exist post-antisecretory treatment.

Aim of the present study is to investigate the effect of therapy with esomeprazole or rabeprazole on the mechanism of pathogenesis of gastritis and particularly on the pattern of release of pro- and anti- inflammatory cytokines associated to peptic ulcerative process by the gastric mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Abdominal pain or discomfort and/or
* Epigastric pain with nausea and vomiting and/or
* Dyspepsia.

Exclusion Criteria:

* Recent upper GI bleeding
* Gastric carcinoma
* Diabetes mellitus
* Liver cirrhosis
* Acute or chronic renal failure
* The ingestion of any antimicrobial or antisecretory medication for at least 15 days prior to endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on changes of cytokines levels in serum of patients | Baseline and 8 weeks

SECONDARY OUTCOMES:
Effect of treatment on changes of cytokines levels in supernatants of cultures of gastric mucosa | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J. Giamarellos-Bourboulis, MD, PhD, Study Chair — 4th Department of Internal Medicine, ATTIKON University Hospital, 124 62 Athens, Greece; Vassileios Koussoulas, MD, PhD, Principal Investigator — Department of Endoscopy, Sismanoglion General Hospital, 151 26 Athens, Greece
Locations (1):
- Department of Endoscopy, Sismanoglion General Hospital, Athens, Greece

REFERENCES:
- [Background] Tzivras M, Koussoulas V, Giamarellos-Bourboulis EJ, Tzivras D, Tsaganos T, Koutoukas P, Giamarellou H, Archimandritis A. Role of soluble triggering receptor expressed on myeloid cells in inflammatory bowel disease. World J Gastroenterol. 2006 Jun 7;12(21):3416-9. doi: 10.3748/wjg.v12.i21.3416. PMID 16733861
- [Background] Koussoulas V, Vassiliou S, Demonakou M, Tassias G, Giamarellos-Bourboulis EJ, Mouktaroudi M, Giamarellou H, Barbatzas C. Soluble triggering receptor expressed on myeloid cells (sTREM-1): a new mediator involved in the pathogenesis of peptic ulcer disease. Eur J Gastroenterol Hepatol. 2006 Apr;18(4):375-9. doi: 10.1097/00042737-200604000-00010. PMID 16538108
- [Derived] Koussoulas V, Giamarellos-Bourboulis EJ, Barbatzas C, Pimentel M. Serum sTREM-1 as a surrogate marker of treatment outcome in patients with peptic ulcer disease. Dig Dis Sci. 2011 Dec;56(12):3590-5. doi: 10.1007/s10620-011-1761-4. Epub 2011 Jun 2. PMID 21633832